CLINICAL TRIAL: NCT01129141
Title: Telehealth Tinnitus Intervention for Patients With TBI
Brief Title: Telephone Tinnitus Education for Patients With Traumatic Brain Injury (TBI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C7452-I
Record Dates: First submitted 2010-05-20; First posted 2010-05-24 (Estimated); Results first posted 2016-11-23 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2016-11

CONDITIONS: Tinnitus
Keywords: Tinnitus; Traumatic Brain Injury Counseling; Counseling; Education; Evaluation studies; Quality of health care
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tele-PTM (Experimental): Telephone-based Progressive Tinnitus Management (Tele-PTM) is a novel home-based telehealth program that involves a series of seven telephone appointments, conducted at approximately 1, 2, 3, 4, and 5 weeks, and 3 and 6 months after enrollment is finalized. Telephone education was provided by the Study Psychologist at weeks 1, 3, and 5, and month 6; and by the Study Audiologist at weeks 2 and 4, and month 3.
  Interventions: Procedure: Tele-PTM
- Wait List Control (Other): Wait List Control subjects received Tele-PTM after completing the 6-month questionnaires. Participants assigned to Wait List Control were instructed that they could receive any available tinnitus services, and that they would receive Tele-PTM following completion of the 3- and 6-month questionnaires.
  Interventions: Procedure: Wait List Control

INTERVENTIONS:
Procedure: Tele-PTM — Telephone-based Progressive Tinnitus Management (Tele-PTM) is a novel home-based telehealth program that involves a series of seven telephone appointments, conducted at approximately 1, 2, 3, 4, and 5 weeks, and 3 and 6 months after enrollment is finalized. Telephone education was provided by the Study Psychologist at weeks 1, 3, and 5, and month 6; and by the Study Audiologist at weeks 2 and 4, and month 3.
  Arms: Tele-PTM
Procedure: Wait List Control — Wait List Control subjects received Tele-PTM after completing the 6-month questionnaires. Participants assigned to Wait List Control were instructed that they could receive any available tinnitus services, and that they would receive Tele-PTM following completion of the 3- and 6-month questionnaires.
  Arms: Wait List Control

SUMMARY:
This study continues the investigators' efforts to develop tinnitus management protocols for Veterans. More specifically, this study developed and evaluated an adaptation of Progressive Tinnitus Management (PTM) for use as a telephone-based program for Veterans and military personnel who have experienced TBI. This adaptation, called Tele-PTM, is a telephone-based program and has the potential of providing needed tinnitus services to Veterans with and without TBI for a relatively small cost and with minimal impact on individual VA hospitals.

DETAILED DESCRIPTION:
Traumatic brain injury (TBI) is strongly associated with tinnitus. Tinnitus management for Veterans and military members with TBI has become a critical concern. The investigators' research has focused on developing effective, evidence-based methods of tinnitus management for Veterans. These efforts led to the development of Progressive Tinnitus Management (PTM). The investigators completed a pilot study to adapt PTM to meet the unique tinnitus management needs of Veterans and military members with TBI using a novel home-based telehealth program called Tele-PTM. Preliminary data analyses indicated that Tele-PTM is effective. The present study modified the PTM program in accordance with pilot study findings and evaluated Tele-PTM using a randomized clinical trial design.

The 4-year study was based at the VA National Center for Rehabilitative Auditory Research (NCRAR). Tele-PTM was implemented and evaluated in a randomized clinical trial. Qualified candidates were randomized to receive either Tele-PTM or Wait-List Control (WLC). All subjects completed questionnaires at baseline and at 3, 6, 9, and 12 months post-baseline. The WLC group received Tele-PTM after completing the 6-month questionnaires. The primary outcome measure was the Tinnitus Functional Index (TFI).

Tele-PTM involves a series of seven telephone appointments, conducted at approximately 1, 2, 3, 4, and 5 weeks, and 3 and 6 months after enrollment is finalized. Telephone education was provided by the Study Psychologist at weeks 1, 3, and 5, and month 6; and by the Study Audiologist at weeks 2 and 4, and month 3.

Tele-PTM has the potential of providing needed tinnitus services to Veterans and active military personnel across the country for a relatively small cost and with minimal impact on individual VA hospitals.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria include:

* "clinically significant" tinnitus according to the initial score on the Tinnitus and Hearing Survey (THS) (minimum total score of 4 on section A; if score is 4-6, one item must be at least 3);
* demonstrates understanding of the requirements of the study (based on adequate responses to the questions by the RC that assess capacity-to-consent);
* has had a hearing test within the past 2 years (and was fitted with hearing aids if appropriate); and
* motivated and capable of participating (including ability to communicate over the telephone in English).

Exclusion Criteria:

* Callers who do not meet all of these criteria will be excluded from study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2011-01; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James A. Henry, PhD, Principal Investigator — VA Portland Health Care System, Portland, OR
Locations (1):
- VA Portland Health Care System, Portland, OR, Portland, Oregon, United States

REFERENCES:
- [Result] Henry JA, Griest S, Thielman E, McMillan G, Kaelin C, Carlson KF. Tinnitus Functional Index: Development, validation, outcomes research, and clinical application. Hear Res. 2016 Apr;334:58-64. doi: 10.1016/j.heares.2015.06.004. Epub 2015 Jun 12. PMID 26074306
- [Derived] Henry JA, Thielman EJ, Zaugg TL, Kaelin C, McMillan GP, Schmidt CJ, Myers PJ, Carlson KF. Telephone-Based Progressive Tinnitus Management for Persons With and Without Traumatic Brain Injury: A Randomized Controlled Trial. Ear Hear. 2019 Mar/Apr;40(2):227-242. doi: 10.1097/AUD.0000000000000609. PMID 29847413

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Potential participants (candidates) were referred to the study by fliers posted at U.S. VA and Military sites. Civilians were not actively recruited for the study, but some discovered it via clinicaltrials.gov or by word of mouth. Candidates contacted the study team and were screened for potential eligibility over the phone.
Pre-assignment Details: Candidates must have had a hearing test within the previous 2 years. They were required to get hearing aids if recommended and wear them for at least 1 month before entering the study. Consented candidates were assessed for phone counseling suitability. If current suicidal ideation (SI) was expressed, the subject was excluded from the study.
Period: Overall Study
Arm/Group | Tele-PTM | Wait List Control
Started | 101 | 104
Completed | 86 | 91
Not Completed | 15 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tele-PTM | Wait List Control | Total
Number analyzed (Participants) | 101 | 104 | 205
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 65 | 73 | 138
  >=65 years | 36 | 31 | 67
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.24 (10.18) | 57.92 (10.71) | 59.07 (10.49)
Gender [Count of Participants; unit: Participants]
  Female | 14 | 16 | 30
  Male | 87 | 88 | 175
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 101 | 104 | 205

OUTCOME MEASURES:

1. Primary Outcome: Tinnitus Functional Index
Description: The TFI served as the primary outcome measure. The TFI is a 25-item self-report questionnaire that has documented validity both for scaling the severity and negative impact of tinnitus, and for measuring treatment-related changes in tinnitus (responsiveness) (Meikle et al., 2012). The total score for the TFI ranges from 0 to 100, with higher scores indicating greater problems with tinnitus. The TFI has excellent internal consistency (Cronbach's α = .97) and high test-retest reliability (r = .86) (Meikle et al., 2012). The authors of the TFI estimated that a 13-point decrease on the TFI for an individual is likely to reflect a change that feels meaningful to the person.
Time Frame: Baseline, 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tele-PTM | Wait List Control
Number analyzed (Participants) | 101 | 104
units on a scale
  Baseline | 69.9 (15.3) | 68.2 (18.7)
  6 months | 47.8 (21.8) | 66.8 (18.3)
Statistical Analysis 1: Comparison: Tele-PTM vs Wait List Control; Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = -17.198, 95% CI 2-sided [-22.86 to -11.53], Standard Error of Mean 2.88

ADVERSE EVENTS:
Arm/Group | Tele-PTM | Wait List Control
Serious Adverse Events (participants affected / at risk) | 0/101 | 0/104
Other Adverse Events (participants affected / at risk) | 0/101 | 0/104

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes